CLINICAL TRIAL: NCT01662349
Title: A Single Center, Pilot Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Plasma Treatment System in Treating Back Acne
Brief Title: Safety Study of Plasma Treatment System to Treat Back Acne
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to other research priorities.
Sponsor: Moe Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOE - 121
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

ARMS (1):
- Plasma (Experimental): Plasma applied to back for up to 20 minutes, twice/week for 4 weeks
  Interventions: Device: MOE Antimicrobial Plasma Treatment System

INTERVENTIONS:
Device: MOE Antimicrobial Plasma Treatment System — Plasma applied to back for up to 20 minutes, twice/week for 4 weeks

SUMMARY:
The purpose of this study is to evaluate the safety of treating human skin with atmospheric plasma and get an initial evaluation of the efficacy of this treatment for acne.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-nursing females age 18-40 years old.
2. Presence of clinically-evident back acne.
3. Minimum of 20 non-inflammatory lesions (open and closed comedones)
4. Minimum of 30 total lesions (sum of inflammatory and non-inflammatory)
5. Subject must have measurable sebum production.
6. Subjects must be in generally good health.
7. Must be able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Any nodulo-cystic lesions at Baseline
2. Pregnancy or breast feeding
3. Use of acne devices or systemic therapy with antibiotics within four months prior to start and throughout the duration of the study
4. Intake of any oral retinoids within four months prior to study start and throughout the duration of the study
5. Topical use of topical retinoids within two weeks prior to study start and throughout the duration of the study
6. Topical use of antibiotics, steroids and/or other non-retinoid topical acne products within two weeks prior to study start and throughout the duration of the study
7. Use of an experimental drug or device within 30 days prior to study start;
8. Intake of hormonal therapy within 3 months prior to study start
9. Use of topical products on the back containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non mild cleansers or moisturizers containing retinol, salicylic or α- or β-hydroxy acids.
10. Concomitant use of mega-doses of certain vitamins, such as vitamin D (>2000IU QD) vitamin B12, haloperidol, halogens such as iodide and bromide, lithium, hydantoin and phenobarbital.
11. Procedures on the skin of the back such as chemical or laser peel, microdermabrasion, photodynamic therapy) within the past 2 weeks or during the study.
12. History or evidence of other skin conditions or diseases that may require concurrent therapy or may interfere with the evaluation of the study medication
13. Any significant medical conditions that could confound the interpretation of the study results.
14. History of/or current skin cancer cancer
15. Use of tanning booths, sun lamps within the past 2 weeks or during the study
16. Any metallic implants or prostheses in the vicinity of the treatment site (such as shoulders, back, spine, pacemakers, etc.).
17. Any known photosensitivity disorders felt by the investigators to preclude safe inclusion in the study.
18. History of significant post-inflammatory hyperpigmentation at the sites of acne lesions.
19. History of or is currently immunocompromised.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in number of reported adverse events | Change from Baseline to 1 month post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B. Kimball, MD, Principal Investigator — Partners Healthcare System
Locations (1):
- Clinical Unit for Research Trials and Outcomes in Skin (CURTIS), Boston, Massachusetts, United States